CLINICAL TRIAL: NCT06255730
Title: The Effect of Stellate Ganglion Block on Insomnia Patients: a Pre - and Post Control Experiments
Brief Title: The Effect of Stellate Ganglion Block on Insomnia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGB shimian old
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stellate Ganglion Block Group (Experimental): Stellate Ganglion Block Group will be given Stellate Ganglion Block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g), once a day
  Interventions: Procedure: Stellate Ganglion Block; Drug: Lidocaine Hydrochloride

INTERVENTIONS:
Procedure: Stellate Ganglion Block — the patients in the observation group were provided with Stellate Ganglion Block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate Ganglion Block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
Drug: Lidocaine Hydrochloride — the patients in the observation group were provided with Stellate Ganglion Block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate Ganglion Block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Other Names: Stellate Ganglion Block

SUMMARY:
A prospective study was conducted on Insomnia Patients. All the patients were provided with Stellate Ganglion Block. The quality of sleep was evaluated to see if Stellate Ganglion Block can improve Insomnia.

DETAILED DESCRIPTION:
Insomnia is a sleep disorder characterized by difficulty falling asleep, staying asleep, or experiencing non-restorative sleep, despite having adequate opportunity for sleep. It is a common condition that can significantly impact an individual's quality of life and overall well-being.A prospective study was conducted on Insomnia Patients. All the patients were provided with Stellate Ganglion Block. The quality of sleep was evaluated to see if Stellate Ganglion Block can improve Insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia patients with the ages over 18.
* Meeting the diagnostic criteria for chronic insomnia as per the International Classification of Sleep Disorders (ICSD) or the Diagnostic and Statistical Manual of Mental Disorders (DSM).
* Experiencing insomnia symptoms persistently for at least three months.
* Not currently using or ceased using medication for insomnia for at least four weeks.
* Willing to undergo Stellate Ganglion Block treatment and participate in the study.

Exclusion Criteria:

* Patients with severe cardiovascular disease, pulmonary disease, or other serious physical health issues.
* Pregnant or lactating women.
* Patients with mental disorders (such as major depression, anxiety disorders, schizophrenia, etc.) or cognitive impairments.
* Patients with known allergies or contraindications to Stellate Ganglion Block treatment.
* Patients currently participating in other clinical trials or receiving experimental treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | day 1 and day 10
  Pittsburgh Sleep Quality Index (PSQI): The PSQI is a widely used scale that assesses sleep quality, including aspects such as sleep latency, sleep duration, sleep efficiency, sleep disturbances, and daytime dysfunction. The total score ranges from 0 to 21, with higher scores indicating worse sleep quality.

SECONDARY OUTCOMES:
Anxiety | day 1 and day 10
  The anxiety was assessed using the Generalized Anxiety Disorder-7, including items related to fear, worry, attention, etc. The total score ranged from 0 to 21, which was positively correlated with potential anxiety. In the previous study, the scale demonstrated a Cronbach's α-coefficient of 0.879.
Sleep Impairment Index | day 1 and day 10
  Sleep Impairment Index (SII): The SII is a scale that measures the impact of sleep disorders on daily functioning. It includes nine items, covering aspects such as feeling unwell in the morning and feeling tired during the day. The total score ranges from 0 to 36, with higher scores indicating more severe sleep impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Chair — Site Coordinator of United Medical Group
Locations (1):
- Center Rehabilitation Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No